CLINICAL TRIAL: NCT01933243
Title: Treatment of Anxiety and Anorexia Nervosa in Adolescents
Acronym: TAANA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrea Bonny (Other)
Responsible Party: Sponsor-Investigator, Andrea Bonny, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAANA-287112
Record Dates: First submitted 2013-08-09; First posted 2013-09-02 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Anxiety; Anorexia Nervosa
Keywords: Anxiety; Anorexia nervosa; Adolescents; Fish oil
MeSH Terms: conditions — Anxiety Disorders; Anorexia Nervosa | interventions — Fish Oils; Eicosapentaenoic Acid; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish oil (Experimental): Fish oil for 12 weeks
  Interventions: Drug: Fish oil
- Placebo pill (Placebo Comparator): Placebo pills for 12 weeks
  Interventions: Drug: Placebo pill

INTERVENTIONS:
Drug: Fish oil — Participants will take 4 capsules daily
  Other Names: ProEPA Xtra soft gel capsules; Eicosapentaenoic acid (2120mg)/ docosahexaenoic acid (600mg)
  Arms: Fish oil
Drug: Placebo pill — Participants will take 4 capsules daily
  Other Names: soybean oil placebo capsules
  Arms: Placebo pill

SUMMARY:
Adolescents with anorexia nervosa frequently have associated anxiety, and standard medications used for anxiety are unhelpful when patients are malnourished. This is a 12 week trial examining the safety, tolerability, and effectiveness of fish oil nutritional supplements for anxiety in adolescents with anorexia nervosa.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is an eating disorder characterized by a morbid fear of weight gain and a perception of being overweight despite objective evidence of weight loss and malnutrition. It has been estimated that almost 0.9% of women will suffer from AN at some point in their lives, and most cases of AN arise during adolescence. Even with appropriate treatment, only about half of patients with AN will have a full recovery, 30% partial recovery, and 20% will progress to having a chronic illness. Earlier, more aggressive treatment with appropriate nutritional recovery during adolescence offers the best chance of a full recovery. Treatment of AN is complicated by the high rate of comorbid psychiatric diagnoses, the physical and cognitive effects of the attendant malnutrition, and the lack of effective pharmacologic interventions. Approximately 75% of patients with AN have a comorbid psychiatric illness, including depression, obsessive compulsive disorder, and anxiety. Anxiety disorders in particular share attributes with AN, including perfectionism, rigidity, compulsivity, and harm avoidance in addition to trait anxiety. Complicating treatment, the risk and severity of patients' anxiety is enhanced by a lower body mass index (BMI), and this low BMI is the likely reason why standard medication treatments for generalized anxiety, such as selective serotonin reuptake inhibitors are ineffective. In order to address these treatment challenges, we propose to study the tolerability, feasibility and efficacy of a non-pharmacologic interventions for anxiety in adolescents with AN: omega-3 polyunsaturated fatty acid (PUFA) supplementation.

Over the past 15 years, there has been an interest in possible associations between fish oil and affective illness, particularly depression. Low plasma levels of docosahexaenoic acid, an essential fatty acid found in fish oil, are associated with low concentrations of cerebrospinal fluid 5-hydroxyindolacetic acid (5-HIAA), a marker of central nervous system serotonin turnover. Epidemiologically, those populations with higher fish oil consumption tend to have lower rates of depression, and reported low levels of fish consumption have been associated with a greater risk of depression in women. It has been hypothesized that omega-3 PUFAs alter brain phospholipid composition and enhance membrane fluidity, and this is supported by evidence that supplementation with omega-3 PUFAs decreases brain water proton transverse relaxation times in patients with bipolar disorder. The association with depression and the proposed mechanism of action elicited some interest regarding associations between omega-3 PUFAs and anxiety disorders. Supplementation trials have shown mixed results, with no effects for obsessive compulsive disorder in patients taking maximum doses of selective serotonin reuptake inhibitors, and another showing decreased anxiety symptoms in 22 patients enrolled in a substance abuse treatment program. Recently, Kiecolt-Glaser and colleagues described a decrease in test-related anxiety symptoms in a non-clinical sample of medical students related to supplementation with omega-3 PUFAs. Although there has been some interest in the use of omega-3 PUFA supplementation as an adjunctive treatment for anorexia nervosa, there have been no systematic trials.

ELIGIBILITY:
Inclusion Criteria:

Females admitted to Nationwide Children's Hospital Eating Disorder Partial Hospitalization Program

Exclusion Criteria:

1. Inability to take pills
2. Co-morbid medical conditions affecting appetite and weight (e.g., inflammatory bowel disease, cancer, cystic fibrosis)
3. Co-morbid psychiatric conditions affecting appetite and weight (e.g., bipolar disorder, substance abuse)
4. Currently taking fish oil supplements
5. Inability to participate in study for 12 consecutive weeks.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2013-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bonny, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PUFA: Fish oil for 12 weeks
  Fish oil: Participants will take 4 capsules daily
Period: Overall Study
Arm/Group | PUFA | Placebo Pill
Started | 12 | 12
Completed | 10 | 8
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- PUFA: Participants randomized to omega-3 PUFA
- Placebo: Participants randomized to placebo
- Total: Total of all reporting groups
Arm/Group | PUFA | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (1.3) | 14.4 (1.8) | 14.7 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 19.6 (2.0) | 18.8 (2.1) | 19.2 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Medication Side Effects Score
Description: At 6 and 12 weeks, medication tolerability was assessed via self-report of nine potential side effects (e.g. diarrhea, burping). Participants were asked whether they experienced these side effects "never, rarely, occasionally, frequently, or very frequently." Individual responses were assigned a numeric equivalent from 0 to 4, and summed for a total side effect score ranging from 0 to 36. Higher scores indicated greater frequency of side effects and lower medication tolerability.
Time Frame: 6 and12 weeks
Population: Participants who completed at least a baseline study visit.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | PUFA | Placebo
Number analyzed (Participants) | 12 | 12
Score on a scale
  6 Weeks: number analyzed (Participants) | 12 | 10
  6 Weeks | 9.5 (1.7) | 6.2 (2.0)
  12 Weeks: number analyzed (Participants) | 10 | 8
  12 Weeks | 6.4 (1.8) | 4.1 (2.0)

2. Secondary Outcome: Beck Anxiety Inventory-Trait (BAIT)
Description: The BAIT is a 21-item self-report measure of anxiety severity rated on a 4-point Likert scale (0= rarely or never; 3= almost always). It has shown acceptable reliability and validity in an adolescent psychiatric inpatient population. BAIT scores over 26 indicate severe anxiety, scores 16-25 indicate moderate anxiety, scores 8-15 indicate mild anxiety, and scores 0-7 indicate a minimal level of anxiety. We chose to measure trait anxiety to examine beyond meal-related (state) anxiety.
Time Frame: Baseline, 6 weeks, and 12 weeks
Population: All participants who completed a baseline study visit
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | PUFA | Placebo
Number analyzed (Participants) | 12 | 12
Score on a scale
  Baseline | 26.4 (2.8) | 19.3 (3.0)
  6 Weeks: number analyzed (Participants) | 12 | 10
  6 Weeks | 21.9 (2.8) | 11 (3.0)
  12 Weeks: number analyzed (Participants) | 10 | 8
  12 Weeks | 14.9 (3.0) | 6.5 (3.3)

3. Other Pre Specified Outcome: Number of Participant Tolerating Saliva Collection and 24 Hour Heart Rate Monitor Use
Description: At baseline, 6 weeks, and 12 weeks, study participants were asked to collect salivary samples 5 times over a 24 hour period. In addition, participants were asked to wear a 24 hour heart monitor during this same 24 hour interval. Compliance wtth completion of these physiological measures was assessed as follows:
  1. For saliva collection, compliance was assessed by return of 5 full vials of saliva with record of time collected.
  2. For 24 hour heart rate monitor, compliance was assessed by return of monitor with then downloading of data to confirm that the participant wore the device during the specified time interval.
Time Frame: Baseline, 6 weeks, and 12 weeks
Population: All participants completing at least a baseline visit.
Measure: Count of Participants; unit: Participants
Arm/Group | PUFA | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Tolerated Saliva Collection | 12 | 12
  Tolerated 24 Hour Heart Rate Monitor | 12 | 12

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | PUFA | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/12 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PUFA (N=12) | Placebo (N=12)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Rash from EKG lead
Suidical Ideation (Psychiatric disorders) | 2 (2) | 1 (1)
Swelling of Eyelid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study limitations include small sample size and reliance on self-reported medication adherence.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No